CLINICAL TRIAL: NCT01207102
Title: A Phase II Study of Abraxane® and Carboplatin as First-line Treatment for "Triple Negative" (Demonstrating no Expression for Estrogen, Progesterone, or Human Epidermal Growth Factor Receptor 2 (HER2)Receptors) Metastatic Breast Cancer
Brief Title: Study Of Abraxane® And Carboplatin As First-Line Treatment For Triple Negative Metastatic Breast Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Low enrollment and there is insufficient data to publish.
Sponsor: Duke University (Other)
Collaborators: Celgene Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Pro00019321
Record Dates: First submitted 2010-09-10; First posted 2010-09-22 (Estimated); Results first posted 2014-12-15 (Estimated); Last update posted 2014-12-15 (Estimated); Status verified 2014-08

CONDITIONS: Metastatic Breast Cancer
Keywords: Breast cancer; Triple negative
MeSH Terms: conditions — Breast Neoplasms | interventions — Albumin-Bound Paclitaxel; Carboplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Abraxane, Carboplatin (Experimental): Abraxane 100mg/m2 IV days 1, 8 and 15 of a 28 day cycle Carboplatin area under the concentration curve, (AUC)2 IV days 1,8, and 15 of a 28 day Cycle
  Interventions: Drug: Abraxane; Drug: Carboplatin

INTERVENTIONS:
Drug: Abraxane — Abraxane® 100 mg/m2 IV over 30 min days 1,8,15 every 28 days
  Other Names: paclitaxel protein-bound particles for injectable suspension
Drug: Carboplatin — area under curve(AUC)=2 over 15 minutes days 1,8,15 every 28 days
  Other Names: Paraplatin

SUMMARY:
Taxanes (such as paclitaxel) are highly active to treat breast cancer. Abraxane® (nanoparticle albumin-bound paclitaxel) compared to standard paclitaxel improves efficacy and tolerability. When combined with a taxane, platinum agents improve response in metastatic breast cancer, with carboplatin conferring less toxicity than cisplatin. The investigators hypothesize that the combination of weekly Abraxane® and carboplatin will lengthen time to progression without producing intolerable toxicity.

DETAILED DESCRIPTION:
Paclitaxel and cisplatin are well-recognized for their activity in treating a variety of tumors including breast cancer. As cytotoxins, they have been studied alone and in combination with other chemotherapeutic agents, and have been incorporated into treatment regimens for women who fail previous anthracycline-based therapies. Although both agents are notable for favorable response rates, they are also associated with a variety of adverse events, some of which may be dose-limiting and having a negative effect on quality of life: myelosuppression, nausea and vomiting, diarrhea, stomatitis/mucositis, short- and long-term neuropathy, nephrotoxicity, alopecia and hypersensitivity reactions.

As second-generation compounds, Abraxane® and carboplatin have been shown to improve response rates and may mediate some of the toxicities associated with paclitaxel and cisplatin, respectively. Of particular interest is Abraxane's potential to reduce allergic reactions associated with other taxanes.

This study combines these two agents: primarily, to evaluate progression-free survival; and secondarily, to assess the feasibility and tolerability of this regimen to treat poor prognosis metastatic breast cancer patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients with histologically or cytologically confirmed diagnosis of metastatic (Stage IV) breast cancer;
* Measurable disease according to Response Evaluation Criteria in Solid Tumors (RECIST);
* "Triple negative" disease defined as "tumor demonstrating no expression for estrogen, progesterone or HER2 receptors." (No expression is categorized as ≤ 10% of cells staining or Allred ≤ 2);
* Aged 18 years or older;
* Eastern Cooperative Oncology Group (ECOG)ECOG/Zubrod performance status of 0 or 1; life expectancy ≥ 3 months;
* No prior chemotherapy for metastatic disease.
* At least 6 months must have elapsed since prior adjuvant chemotherapy.
* Laboratory tests performed within 14 days of study entry showing:

  * Granulocytes ≥ 1,500/µL;
  * Platelets ≥ 100,000/µL;
  * Hemoglobin ≥ 9.0 gm/dL;
  * Total bilirubin ≤ institutional upper limit of normal (ULN);
  * Aspartate transaminase (AST) and alanine aminotransferase (ALT) ≤ 2.5 times ULN;
  * Alkaline phosphatase ≤ 5 times ULN;
  * Estimated creatinine clearance ≥ 60 mL/min.
  * Urine protein:creatinine ratio ≤ 1.0. or 24 hour urine protein collection demonstrating ≤ 1 gram of protein per 24 hours to be eligible.
* left ventricular ejection fraction (LVEF) ≥ 50% by multiple gated acquisition scan (MUGA)/Echocardiogram;
* Informed consent to receive protocol treatment:
* Cognitive and communication skills adequate to comply with study and/or follow-up procedures;
* Geographic proximity and ability to comply with weekly study visits for the duration of the treatment;
* No reproductive potential:

  * If pre-menopausal - Negative serum pregnancy test within 3 days prior to initiation of protocol-based treatment and patient agrees to use contraceptive method (abstinence, intrauterine device, barrier device with spermicide or surgical sterilization) during and for 3 months after completion of protocol treatment;
  * If post-menopausal - Amenorrhea for ≥ 12 months or follicle stimulating hormone (FSH) within post menopausal range.

Exclusion Criteria:

* Pregnant or breast feeding.
* Prior treatment with Abraxane® or carboplatin.
* Prior chemotherapy for metastatic breast cancer.
* Known hypersensitivity to any component of any study drug.
* Active infection.
* Current neuropathy ≥ grade 2.
* central nervous system (CNS) metastases as determined by head CT with contrast or head MRI.
* Uncontrolled congestive heart failure (CHF), or history of myocardial ischemia (MI), unstable angina, stroke, or transient ischemia within previous 6 months.
* Uncontrolled serious contraindicated medical condition or illness.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2011-08; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kimberly L Blackwell, MD, Study Chair — Duke University
Locations (2):
- Duke University Medical Center, Durham, North Carolina, United States
- Peking University School of Oncology/Beijing Cancer Hospital, Beijing, China

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Abraxane, Carboplatin
Started | 10
Completed | 0
Not Completed | 10
Not completed — Withdrawal by Subject | 5
Not completed — Adverse Event | 2
Not completed — progression | 2
Not completed — Withdrawal by Treating Physician | 1

BASELINE CHARACTERISTICS:
Arm/Group | Abraxane, Carboplatin
Number analyzed (Participants) | 10
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 9
  >=65 years | 1
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.5 (8.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10
  Male | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 7
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 2
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 3
  China | 7

OUTCOME MEASURES:

1. Primary Outcome: PFS
Description: The primary objective of the trial is to statistically test whether Abraxane® and carboplatin can improve progression-free survival (PFS) as compared to historical controls.
Time Frame: PFS is defined as the interval from study registration to disease progression or death due to any cause, whichever comes first
Population: Due to insufficient accrual, data analysis was not performed.
Arm/Group | Abraxane, Carboplatin
Number analyzed (Participants) | 0

2. Secondary Outcome: To Assess the Safety and Tolerability of a Combination Regimen of Weekly Abraxane® and Carboplatin to Treat Women With "Triple Negative" Stage IV Metastatic Breast Cancer
Description: The proportion of patients experiencing any neurotoxicity will be tabulated by grade. The proportion of patients experiencing ≥ grade 3 non-hematologic toxicities (excluding neurotoxicity) and the proportion of patients experiencing ≥ grade 3 hematologic toxicities will be calculated with their exact 80% confidence intervals.
Time Frame: 2 years
Population: Due to insufficient accrual, data analysis was not performed.
Arm/Group | Abraxane, Carboplatin
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Arm/Group | Abraxane, Carboplatin
Serious Adverse Events (participants affected / at risk) | 6/10
Other Adverse Events (participants affected / at risk) | 10/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Abraxane, Carboplatin (N=10)
Anemia (Blood and lymphatic system disorders) | 4
Vomiting (Gastrointestinal disorders) | 1
Allergic reaction (Immune system disorders) | 1
Neutrophil count decreased (Investigations) | 5
Platelet count decreased (Investigations) | 1
White blood cell decreased (Investigations) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Abraxane, Carboplatin (N=10)
Anemia (Blood and lymphatic system disorders) | 6
Blood and lymphatic system disorders - Other, specify: lymphedema (Blood and lymphatic system disorders) | 1
Ventricular tachycardia (Cardiac disorders) | 1
Eye disorders - Other, specify: floaters (Eye disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 1
Constipation (Gastrointestinal disorders) | 1
Diarrhea (Gastrointestinal disorders) | 2
Gastritis (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 6
Vomiting (Gastrointestinal disorders) | 5
Chills (General disorders) | 1
Edema limbs (General disorders) | 4
Fatigue (General disorders) | 3
Fever (General disorders) | 1
General disorders and administration site conditions - Other, specify: cold intolerance (General disorders) | 1
Non-cardiac chest pain (General disorders) | 1
Pain (General disorders) | 2
Allergic reaction (Immune system disorders) | 2
Infections -Other: Infection with Grade 3 or 4 neutrophils (ANC <1.0 x 10e9/L) (Infections and infestations) | 1
Sinusitis (Infections and infestations) | 1
Vaginal infection (Infections and infestations) | 1
Alanine aminotransferase increased (Investigations) | 4
Aspartate aminotransferase increased (Investigations) | 3
Neutrophil count decreased (Investigations) | 9
Platelet count decreased (Investigations) | 4
White blood cell decreased (Investigations) | 2
Back pain (Musculoskeletal and connective tissue disorders) | 3
Musculoskeletal and connective tissue disorder - Other, specify: toes stiff upon standing (Musculoskeletal and connective tissue disorders) | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1
Dizziness (Nervous system disorders) | 1
Dysgeusia (Nervous system disorders) | 1
Memory impairment (Nervous system disorders) | 1
Peripheral sensory neuropathy (Nervous system disorders) | 3
Anxiety (Psychiatric disorders) | 2
Urinary frequency (Renal and urinary disorders) | 1
Vaginal dryness (Reproductive system and breast disorders) | 1
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 3
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 2
Respiratory, thoracic and mediastinal disorders - Other, specify: yellow sputum (Respiratory, thoracic and mediastinal disorders) | 1
Alopecia (Skin and subcutaneous tissue disorders) | 3
Dry skin (Skin and subcutaneous tissue disorders) | 1
Nail loss (Skin and subcutaneous tissue disorders) | 1
Urticaria (Skin and subcutaneous tissue disorders) | 1
Flushing (Vascular disorders) | 1
Hot flashes (Vascular disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes